CLINICAL TRIAL: NCT04299074
Title: The Effect of Smartphone Addiction on Physical Activity Level
Brief Title: Smartphone Addiction and Physical Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Meryem BUKE, Principal Investigator, Pamukkale University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 60116787-020/1323
Record Dates: First submitted 2020-02-26; First posted 2020-03-06 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-03

CONDITIONS: Sports Physical Therapy
Keywords: Addiction; Healthy individuals; Physical activity; Smartphone; Sport science
MeSH Terms: conditions — Behavior, Addictive; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Addiction (Other): problematic addiction
  Interventions: Other: addiction

INTERVENTIONS:
Other: addiction — questionnaire

SUMMARY:
This study aimed to determine the effect of smartphone addiction on physical activity level in healthy individuals. A total of 300 (134 female) healthy university students were included in this study. The mean age of the subjects was 21.36 ± 2.33 year.

DETAILED DESCRIPTION:
This study aimed to determine the effect of smartphone addiction on physical activity level in healthy individuals. A total of 300 (134 female) healthy university students were included in this study. The mean age of the subjects was 21.36 ± 2.33 year. The universe of the study consisted of volunteer students (Coaching Education, Physical Education and Sports Teaching, Sports Management, Recreation Departments) at the Faculty of Sport Sciences. Participants' demographic information was obtained and their physical activity levels were questioned with International Physical Activity Questionnaires (IPAQ) and smartphone addictions with the Smartphone Addiction Scale- Short Verison (SAS-SV).

ELIGIBILITY:
Inclusion Criteria:

* to be 18-35 old years

Exclusion Criteria:

* not to be sports science students

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2019-02-20 (Actual); Primary Completion 2019-03-20 (Actual); Study Completion 2019-10-20 (Actual)

PRIMARY OUTCOMES:
Questionnaire | This questionnaire is used during baseline assessment
  International Physical Activity Questionnaires: The higher score obtained from this questionnaire indicated that participant have a high physical activity level. Physically inactive (<600 MET-min / week), low level of physical activity (600 - 3000 MET minutes / week) and the adequate level of physical activity (beneficial to health) (> 3000 MET minutes / week).
Scale | This scale is used during baseline assessment
  Smartphone Addiction Scale- Short Verison: The higher score obtained from this scale indicated that participant have smartphone addiction. Cut-off score was 31 for male and 33 for female

CONTACTS AND LOCATIONS:
Overall Officials: Meryem BUKE, Principal Investigator — Pamukkale University
Locations (1):
- Pamukkale University, Denizli, Kinikli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No